CLINICAL TRIAL: NCT02053402
Title: Effect of Vitamin d Supplementation on the Control of Persistent Asthma in Children at Dr George Mukhari Academic Hospital, Pretoria, South Africa
Brief Title: Effect of Vitamin D Supplementation on the Control of Asthma in Children at a South African Academic Hospital
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Limpopo (Other)
Responsible Party: Principal Investigator, Siyazi Mda, Research project supervisor, University of Limpopo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MREC/M/82/2013:PG
Record Dates: First submitted 2014-01-21; First posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Persistent Asthma
Keywords: vitamin D supplementation, persistent asthma, control
MeSH Terms: interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo to be given daily for six months
- Vitamin D (Active Comparator): 1200 IU of vitamin D, daily for six months
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D daily for six months
  Other Names: Cholecalciferol
  Arms: Vitamin D

SUMMARY:
The aim of this randomized double-blind placebo controlled study is to assess whether vitamin D supplementation will improve control in South African children with persistent asthma at an academic hospital.

The following hypotheses will be tested: Vitamin D significantly and directly correlates with poor control of persistent asthma; Daily vitamin D supplementation for six months will result in improved control of persistent asthma compared to a placebo.

It is intended to enroll 100 children between the ages of 6 to 12 years with persistent asthma on inhaled therapy. The sample size calculations are based on the hypothesis that vitamin D supplementation will result in a 25% improvement in asthma symptoms as measured by the Asthma Treatment Assessment Questionnaire (ATAQ) and peak flow readings. The children will be randomized into one of two groups; one group will be given 1200 IU of vitamin and the other a placebo. The vitamin D or placebo will be given in the morning daily to each child for six months. The children will be assessed monthly by the study physician, to evaluate for signs of poor asthma control e.g. persistent cough and recurrent wheezing. The heights and weights and peak expiratory flow meter readings will also be obtained monthly for six months. Blood samples will be taken for Vitamin D levels, calcium, phosphorus levels at baseline, third month and at the end of the study. All enrolled children will be required to produce their tablet containers for pill counting on a monthly basis to ensure adherence.

DETAILED DESCRIPTION:
Some studies have demonstrated a link between Vitamin D deficiency and poor asthma control. Vitamin D has been shown to have an immune modulatory role and plays a role in improving the response to corticosteroids which are the mainstay of treatment in persistent asthma.

A randomized double-blind placebo controlled study will be performed to assess whether vitamin D supplementation will improve control in South African children with persistent asthma at an academic hospital.

The researchers intend to enroll 100 children between the ages of 6 to 12 years with persistent asthma on inhaled therapy. The children will be enrolled from the pediatric outpatient department of Dr George Mukhari Academic Hospital, which is in Pretoria, South Africa. After enrolment, the children will be randomized into one of two groups; one group of 50 children will be given 1200 IU of vitamin and the other group of 50 will receive a placebo. The sample size calculations are based on the hypothesis that vitamin D supplementation will result in a 25% improvement in asthma symptoms as measured by the Asthma Treatment Assessment Questionnaire (ATAQ) and peak flow readings.

The following groups of children will be excluded: children with intermittent asthma symptoms; children whose caregivers refuse to give signed informed consent; children who are not able to use a peak expiratory flow meter and those with concomitant chronic respiratory and/or cardiac conditions.

The vitamin D or placebo will be given in the morning daily to each child for six months. The date when the child was first diagnosed as having asthma will be noted, as well as the date of asthma treatment initiation, and the current treatment at enrolment will be recorded. The children will be asked to come to the hospital for follow up at monthly intervals. At these monthly visits, the children will be evaluated for signs and symptoms of poor asthma control by the study physician. The heights and weights of the children will be measured and peak expiratory flow meter readings will also be obtained monthly for six months. Blood samples will be taken for Vitamin D levels, calcium, phosphorus levels at baseline, third month and at the end of the study. Treatment adherence will be assessed by counting the pills in the containers by the study physician at the monthly visits. All enrolled children will be required to produce their tablet containers for pill counting.

Data will be analyzed using the IBM SPSS Statistics program. Analysis of variance will be performed in order to compare the difference in ATAQ scores and peak flow meter reading from baseline to six months post intervention between the two groups (vitamin D and placebo).

ELIGIBILITY:
Inclusion Criteria:

- Children aged 6 to 12 years with persistent asthma on inhaled therapy, attending the pediatric outpatient department at Dr George Mukhari Academic Hospital in Pretoria, South Africa.

Exclusion Criteria:

- Children with intermittent asthma; Children whose caregivers refuse to give signed informed consent; Children who are not able to use a peak expiratory flow meter and those with a concomitant chronic respiratory and/or cardiac condition

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-01 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in peak flow meter reading from baseline to six months, between vitamin D and placebo groups | From "Day 1" up to until six months of supplementation
  Children will be assessed monthly for control of persistent asthma by peak flow meter readings.The peak flow meter readings will be obtained monthly, from each child for six months. The difference in the peak flow meter reading from baseline to six months and between the two treatment groups will be assessed.

SECONDARY OUTCOMES:
Assessment of correlation between vitamin D levels and peak flow meter readings and Asthma Treatment Assessment Questionnaire scores. | On day 1
  Vitamin D levels and peak flow meter readings and Asthma Treatment Assessment Questionnaire scores will be obtained at enrolment. The correlation between vitamin D levels and peak flow meter readings will be evaluated. The correlation between vitamin D levels and Asthma Treatment Assessment Questionnaire scores will also be assessed.
Comparison of change from baseline in Asthma Treatment Assessment Questionnaire score at six months, between vitamin D and placebo groups | From Day 1 up to six months of supplementation
  Asthma Treatment Assessment Questionnaire (ATAQ). ATAQ includes questions regarding several aspects of asthma management in addition to asthma control, including satisfaction with patient-provider communication, patient attitudes and behaviors, and perceived self-efficacy. The instrument was designed to assist clinicians and health plans with identifying children with poorly controlled asthma who may be candidates for additional asthma-management support. The ATAQ scores will be obtained monthly for six months. The difference in ATAQ scores from baseline enrolment to six months between the two treatment (vitamin D and placebo) groups will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Siyazi Mda, MBChB, PhD, Study Chair — Univeristy of Limpopo, Medunsa Campus
Locations (1):
- Dr George Mukhari Academic Hospital, Pretoria, Gauteng, South Africa